CLINICAL TRIAL: NCT04338087
Title: The Correlation Between Assisted Reproductive Technology and Male Erectile Dysfunction.
Brief Title: The Effect of Assisted Reproductive Technology on Male Sexual Function.
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0102-17-RMB
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fertility treatments: Men participating in fertility treatments.
  Interventions: Other: Questionnaire and personal interviews.
- Spontaneous pregnancy: Men whose wives conceived spontaneously.
  Interventions: Other: Questionnaire and personal interviews.

INTERVENTIONS:
Other: Questionnaire and personal interviews. — Questionnaire and personal interviews.

SUMMARY:
Men participating in assisted reproductive technology treatments will be recruited to a study involving filling erectile function questionnaires throughout fertility treatments, pregnancy and up to 1 year after birth.

DETAILED DESCRIPTION:
Men participating in fertility will be recruited to a study involving filling erectile function questionnaires throughout fertility treatments, pregnancy and up to 1 year after birth. In addition, participants will be questioned regarding marital life, sexual intercourse frequency, medical history and treatments for erectile dysfunction in relevant cases. Thes control group will be comprised of male subjects who did not require fertility treatments to conceive.

ELIGIBILITY:
Inclusion Criteria:

* Participation in fertility treatments.

Exclusion Criteria:

* None.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Study Population: Male patients participating in fertility treatments.
Sampling Method: Non-Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in International index of erectile function score | From recruitment up to 3 years.
  Changes in International index of erectile function score with a possible score ranging from 0 to 75. The higher the score, the better erectile function is.

SECONDARY OUTCOMES:
Sexual intercourse rate. | From recruitment up to 3 years.
  Sexual intercourse rate as measured by the average monthly intercourse rate.
Use of phospho-di-esterase 5 inhibitors | From recruitment up to 3 years.
  Use of phospho-di-esterase 5 inhibitors as measured by the number of men using this medication.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam healthcare campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No